CLINICAL TRIAL: NCT02310191
Title: Correlation Between Laboratory Markers and Origin of New Brain Ischemic Lesions After Carotid Stenting
Status: Completed | Type: Observational
Sponsor: University Hospital Ostrava (Other)
Responsible Party: Sponsor
Other Study IDs: UHOG-2/2012
Record Dates: First submitted 2014-11-21; First posted 2014-12-08 (Estimated); Last update posted 2014-12-08 (Estimated); Status verified 2014-12

CONDITIONS: Carotid Stenosis; Brain Ischemia; Laboratory Problem
Keywords: ischemic stroke; carotid stenting; MRI diffusion weighted imaging; Laboratory marker
MeSH Terms: conditions — Carotid Stenosis; Brain Ischemia; Ischemic Stroke

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples collecting: hematology + reticulocytes, coagulation markers (PT, APTT, INR, Fbg, Clauss), vWF antigen, PAI-1 activity, PAI-1 polymorphism 4G/g, Multiplate (ASA and clopidogrel resistance test) anti Xa activity
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Stenting: Carotid stenting
  Interventions: Procedure: Carotid stenting

INTERVENTIONS:
Procedure: Carotid stenting — Procedures will be carried out via the femoral approach following a Seldinger technique. All patients will be on long-term aspirin (100 mg/day) and a 525-mg loading dose of clopidogrel. A dose of 10 000 units unfractionated heparin will be administered at the beginning of the intervention. A cerebral protection device (FilterWire EZ™; Boston Scientific, Natick, Massachusetts, USA) will be use in all patients if possible. The type of covered stent and other specific intervention strategies will be left to the discretion of the interventional radiologists. After predilatation of the stenosis (if needed), an appropriate stent for each stenosis will be implanted and then dilated using a balloon catheter.

SUMMARY:
New brain ischemic lesions are detected in about 50% of patients undergoing carotid artery stenting (CAS). The aim was to assess correlation between selected laboratory markers and occurrence of new brain infarctions after CAS.

DETAILED DESCRIPTION:
Methods: All consecutive patients 1) with internal carotid artery stenosis >70%, 2) indicated to CAS, 3) with signed informed consent were enrolled to the prospective study during 16 months. All patients used dual antiplatelet therapy (acetylsalicylic acid [ASA] 100 mg + clopidogrel 75 mg per day) at least 7 days before CAS. Neurological examination and brain magnetic resonance imaging (MRI) were performed before and 24 hours after CAS in all patients. Venous blood samples were collected within 24 hours before CAS in all patients: hematology + reticulocytes, coagulation markers (PT, APTT, INR, Fbg, Clauss), vWF antigen, PAI-1 activity, PAI-1 polymorphism 4G/g, Multiplate (ASA and clopidogrel resistance test). Blood samples for the assessment of anti Xa activity were collected during CAS. T-test was used for statistical evaluation.

ELIGIBILITY:
Inclusion Criteria:

patients

1. With internal carotid artery stenosis >70%
2. Indicated to CAS
3. With signed informed consent. Able to use (acetylsalicylic acid [ASA] 100 mg + clopidogrel 75 mg per day) at least 7 days before CAS

Exclusion Criteria:

* Contraindication for magnetic resonance imaging

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with internal carotid artery stenosis >70%, indicated to carotid stenting
Sampling Method: Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2012-07; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Number of participants with change of level of selected laboratory markers as a measure of potential embolic complication of carotid stenting | blood samples were collected within 24 hours before CAS and anti Xa activity blood samples are collected during CAS procedure
  Laboratory markers:erytrocytes, reticulocyte index, reticulocytes, platelet count, immature platelet fraction, mean platelet volume, prothrombin time (PT), activated parcial tromboplastine time (APTT), international normalized ratio (INR), Fibrinogen (Fbg), Clauss fibrinogen,von Willebrand factor (vWF) antigen, plasminogen activator inhibitor-1 (PAI-1) activity, PAI-1 polymorphism 4G/5G, Multiplate aggregometry , anti Xa activity
Number of participants with correlation of changed level of selected laboratory markers and occurence of new brain ischemic lesion as a measure of safety of carotid stenting procedure | blood samples were collected within 24 hours before CAS and anti Xa activity blood samples are collected during CAS procedure
  Laboratory markers:erytrocytes, reticulocyte index, reticulocytes, platelet count, immature platelet fraction, mean platelet volume, prothrombin time (PT), activated parcial tromboplastine time (APTT), international normalized ratio (INR), Fibrinogen (Fbg), Clauss fibrinogen,von Willebrand factor (vWF) antigen, plasminogen activator inhibitor-1 (PAI-1) activity, PAI-1 polymorphism 4G/5G, Multiplate aggregometry , anti Xa activity

CONTACTS AND LOCATIONS:
Overall Officials: Martin Kuliha, MD, Principal Investigator — University Hospital Ostrava
Locations (1):
- University Hospital Ostrava, Ostrava, Czechia